CLINICAL TRIAL: NCT03102541
Title: Effects of Preoperative High Oral Protein Load on Short- and Long-term Renal Outcomes Following Cardiac Surgery - a Matched Case-control Study
Brief Title: Effects of Oral Protein Load on Kidney Function in Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain, Senior Physician, University of Giessen
Other Study IDs: 79/16 F
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery: 214 adult patients with estimated GFR ≥60 ml/min/1.73 m2 (CKD-Epidemiology Collaboration equation) undergoing elective cardiac surgery (coronary artery bypass, valve replacements, combined or other surgery, with cardiopulmonary bypass) between November 2014 and October 2015 at the San Bortolo Hospital, Vicenza, Italy
  Interventions: Other: None intervention

INTERVENTIONS:
Other: None intervention

SUMMARY:
Acute kidney injury (AKI) occurs in approximately one-third of patients undergoing cardiac surgery (CS), and represents one of the most significant negative predictors of patient outcome in this population. In the healthy adult, a high protein meal is known to enhance glomerular filtration rate and is mediated by an increase in renal blood flow. The investigators hypothesized that preoperative oral protein load may precondition the kidneys for upcoming insults and reduce the rate of postoperative AKI and long-term renal outcome.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) occurs in approximately one-third of patients undergoing cardiac surgery (CS), and represents one of the most significant negative predictors of patient outcome in this population. To date, there is no therapy to prevent AKI. In the healthy adult, a high protein meal is known to enhance glomerular filtration rate (GFR) and is mediated by an increase in renal blood flow. The investigators hypothesized that preoperative oral protein load may induce an adaptive response of the kidneys, and precondition the kidneys for upcoming insults. In the present study, the investigators aimed to compare the prevalence and severity of AKI in patients undergoing oral high protein load of the 'Preoperative Renal Functional Reserve Predict Risk of AKI after Cardiac Operation' study to age- and gender-matched "controls" who had a standard preoperative care the day prior to surgery within the same period (November 2014-October 2015) at San Bortolo Hospital, Vicenza, Italy. Both groups were followed 1 year post-discharge to evaluate long-term renal outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects older than 18 years undergoing elective cardiac surgery
2. Subjects older than 18 years with an estimated eGFR >60 ml/min/1.73 m2 (CKD-EPI)
3. Subjects who signed informed consent forms

Exclusion Criteria:

1. Pregnancy
2. Chronic kidney disease ≥ stage III (KDIGO criteria)
3. Preexisting acute kidney injury (as determined by all available serum creatinine values from hospital and outpatient medical records within the previous 90 days)
4. Solitary kidney
5. Diabetes mellitus type 1
6. Recent cardiac arrest or myocardial infarction up to 7 days before surgery
7. Liver failure or cirrhosis
8. Total parenteral nutrition
9. Haemoglobin <11 g/dl
10. Sepsis
11. History of malabsorption, chronic inflammatory bowel disease, short bowel, or pancreatic insufficiency
12. Transplant donor or recipient
13. Active autoimmune disease with renal involvement
14. Rhabdomyolysis
15. Prostate hypertrophy with International Prostate Symptom Score ≥20
16. Transcatheter aortic valve implantation
17. Active neoplasm
18. Patients who did not pause angiotensin-converting enzyme inhibitors or angiotensin II receptor blockers or received non-steroidal anti-inflammatory drugs a minimum of 48 hours before hospital admission.
19. Patients who received intravenous radiocontrast agents within the 72 hours before hospital admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with estimated GFR ≥60 ml/min/1.73 m2 (CKD-Epidemiology Collaboration equation) undergoing elective cardiac surgery (coronary artery bypass, valve replacements, combined or other surgery, with cardiopulmonary bypass) between November 2014 and October 2015 at the San Bortolo Hospital, Vicenza, Italy
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2016-11-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of AKI after cardiac surgery | 7 days
  using full Kidney Disease: Improving Global Outcomes criteria
Long-term change in estimated GFR | 3 months and 1 year after cardiac surgery
  using CKD-Epidemiology Collaboration creatinine formula

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ronco, MD, Study Director — International Renal Research Institute of Vicenza, Vicenza, Italy

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: SAP
Time Frame: Starting immediately after results have been published
Access Criteria: by email request to first author

REFERENCES:
- [Background] Zarbock A, Schmidt C, Van Aken H, Wempe C, Martens S, Zahn PK, Wolf B, Goebel U, Schwer CI, Rosenberger P, Haeberle H, Gorlich D, Kellum JA, Meersch M; RenalRIPC Investigators. Effect of remote ischemic preconditioning on kidney injury among high-risk patients undergoing cardiac surgery: a randomized clinical trial. JAMA. 2015 Jun 2;313(21):2133-41. doi: 10.1001/jama.2015.4189. PMID 26024502
- [Background] Sharma A, Zaragoza JJ, Villa G, Ribeiro LC, Lu R, Sartori M, Faggiana E, de Cal M, Virzi GM, Corradi V, Brocca A, Husain-Syed F, Brendolan A, Ronco C. Optimizing a kidney stress test to evaluate renal functional reserve. Clin Nephrol. 2016 Jul;86(7):18-26. doi: 10.5414/CN108497. PMID 27285313
- [Derived] Husain-Syed F, Emlet DR, Wilhelm J, Danesi TH, Ferrari F, Bezerra P, Lopez-Giacoman S, Villa G, Tello K, Birk HW, Seeger W, Giavarina D, Salvador L, Fuhrman DY, Kellum JA, Ronco C; IRRIV-AKI Study Group. Effects of preoperative high-oral protein loading on short- and long-term renal outcomes following cardiac surgery: a cohort study. J Transl Med. 2022 May 10;20(1):204. doi: 10.1186/s12967-022-03410-x. PMID 35538495